CLINICAL TRIAL: NCT00158158
Title: Interventions for Tobacco Dependent Adolescents
Brief Title: Effectiveness of Reducing Smoking in Facilitating Smoking Cessation in Adolescents - 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Dorothy Hatsukami, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14538-2; R01-14538-2; DPMC
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
Keywords: smoking addiction
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Usual care
  Interventions: Drug: Usual Care
- 2 (Experimental): Reduction in smoking
  Interventions: Other: Smoking Reduction

INTERVENTIONS:
Drug: Usual Care — If unable to quit at quit date, offered usual care to set another quit date.
  Other Names: Nicoderm used for initial quit attempt.
  Arms: 1
Other: Smoking Reduction — If unable to quit smoking, reduce smoking rate prior to quit date.
  Other Names: Nicotine patch used for initial cessation and smoking reduction.
  Arms: 2

SUMMARY:
Currently one in five high school students smoke. Smoking can harm adolescents well before they reach adulthood by causing a number of immediate, sometimes irreversible, health risks and problems. This study will examine whether reducing smoking will facilitate quitting smoking in adolescents who have unsuccessfully attempted to quit smoking

DETAILED DESCRIPTION:
Among adolescents, the short-term health effects of smoking include damage to the respiratory system, addiction to nicotine, and the associated risk of other drug use. Adolescents are at greater risk for long-term health problems, including several types of cancer. This study will examine whether reducing smoking will facilitate smoking cessation in adolescents who have unsuccessfully attempted to quit smoking. The study will also assess whether reduction of smoking leads to continued involvement in treatment, less toxic cigarette exposure, and improved motivation and self-efficacy to quit.

Participants in this open-label study will undergo 2 weeks of baseline measurements, followed by 2 weeks of smoking cessation treatment. Treatment will involve a nicotine patch, for those who are eligible, and a standardized behavioral intervention aimed at supporting smoking cessation. Those who are ineligible to receive a nicotine patch will only receive the standardized behavioral intervention. Participants who quit smoking during the first phase of treatment will continue to receive the nicotine patches and/or the standardized behavioral intervention. Those who are still smoking after the first treatment will be randomly assigned to one of two conditions and will continue to use nicotine patches for 4 weeks. Group 1 will receive standardized behavioral therapy and will set a specific quit date. Group 2 will be encouraged to decrease smoking by 50% the first week and 75% the second week. During Week 3, participants will be encouraged to completely quit smoking. Study visits will occur weekly, at which time nicotine patches will be dispensed, standardized behavioral therapy will be provided, and standard physiological measurements will be taken. A urine sample will also be collected. Follow-up visits will be held 2 weeks, 3 weeks, and 6 months following completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Has smoked at least 5 cigarettes a day for at least 6 months
* Does not regularly use other tobacco products
* Motivated to quit smoking
* Not currently using medications to quit smoking
* Willing to use an effective form of contraception throughout the study

Exclusion Criteria:

* Informed that nicotine replacement therapy is medically inadvisable
* Diagnosed with a psychiatric disorder within 3 months prior to enrollment
* Currently taking an unstable dose of psychoactive medications
* Currently taking medications that may react with a nicotine patch
* History of alcohol or drug abuse within 3 months prior to enrollment
* Pregnant

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Quit Rate; measured throughout study | 26 weeks
Extent of reduction in smoking; measured at Week 6 | 6, 12 and 26 weeks

SECONDARY OUTCOMES:
Degree of motivation to quit; measured at Week 6 | 6, 12 and 26 weeks
Extent of exposure to cigarette toxicity; measured throughout study | 6, 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States